CLINICAL TRIAL: NCT06558487
Title: The Internal Prospective validatiON of a prediCtiOn Model for the Change of admIssion for Patient With caNcer Admitted to the emerGency Department (ONCOMING Study)
Brief Title: The Internal Prospective Validation of the Cancer Admission Score (CAS) Prediction Model
Acronym: ONCOMING
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jason den Duijn, Principal Investigator, Erasmus Medical Center
Other Study IDs: 12821
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Oncology
Keywords: cancer care; emergency care; prediction model; admission
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer patients: All adult patients with an active cancer diagnosis who visit the emergency department (ED) of the Erasmus University Medical Centre (Erasmus MC).
  Interventions: Other: Cancer Admission Score Prediction Model

INTERVENTIONS:
Other: Cancer Admission Score Prediction Model — A prediction model that calculates the chance for a patient to be admitted after triage and after first blood results

SUMMARY:
The goal of this single center prospective observational study is to determine the agreement between the cancer admission score (CAS) predicted disposition and the actual disposition in patients with an active cancer diagnosis visiting the emergency department (ED). The main question it aims to answer are: Is the performance of the CAS good enough to play a potential role in the ED care process. For each participant the CAS will be calculated and compared to the actual outcome.

DETAILED DESCRIPTION:
The goal of this single center prospective observational study is to determine the agreement between the cancer admission score (CAS) predicted disposition and the actual disposition in patients with an active cancer diagnosis visiting the emergency department (ED). The main question it aims to answer are: Is the performance of the CAS good enough to play a potential role in the ED care process.

The first part of this study is an observational part. For patients with cancer that are presented to the emergency department (ED) the cancer admission score (CAS) will be calculated by the model both after triage and after the first blood results are in. Furthermore, the expected disposition will be asked to the attending nurse after triage and after the first blood results. Finally, the actual disposition will be written down after the patient has left the ED, in combination with ED length of stay (LOS) and the time for the attending physician to reach a decision about the disposition (time-to-disposition) and the time for a patient to leave the ED (time-to-leave).

The second part is the interventional part. In this part we introduce an early bed reservation intervention. The CAS is still calculated for the patient. If the CAS is 80% or higher based on the triage, the attending physician will be alerted and a call to the bed coordinator will be placed to reserve a bed in advance. After the first blood results are known the second CAS will be calculated, if this drops below 70% the reserved bed can be canceled by the attending physician. Similar to the first part, the expected disposition from the attending nurse after triage and after first blood results will be collected. Finally, the actual disposition, ED LOS, time-to-disposition and time-to-leave will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid or hematological malignancies and receiving systemic therapy or having received systemic therapy within the last 3 months.
* Presented at or admitted from the emergency department for the oncology, hematology neuro- or lung-oncology clinical unit.

Exclusion Criteria:

* <18 years old
* Only received a surgical intervention as cancer treatment
* Admitted to the ED for the surgical department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with an active cancer diagnosis who visit the ED of the Erasmus University Medical Center (Erasmus MC).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer Admission Score | Through study completion, an average of 6 months
  Cancer Admission Score (CAS) calculated after triage and after first blood results, ranging from 0 to 100%. The higher the score the greater the change of admission
Disposition | Through study completion, an average of 6 months
  The outcome of a visit to the ED, being either admission or home
Agreement between the CAS and the actual disposition | Through study completion, an average of 6 months
  Agreement between the CAS predicted outcome and the actual outcome

SECONDARY OUTCOMES:
Agreement between expected disposition by nurse and actual disposition | Through study completion, an average of 6 months
  Agreement between the nurse predicted outcome and the actual outcome
time-to-disposition | Through study completion, an average of 6 months
  The average time between patient's arrival at the emergency department (ED) and the decision to disposition
time-to-leave | Through study completion, an average of 6 months
  The average time between the decision to disposition and departure from the ED (either home or ward)
ED Length of Stay | Through study completion, an average of 6 months
  The total time spent in the ED by a patient during their visit

OTHER OUTCOMES:
Sex | Through study completion, an average of 6 months
  The sex of a patient
Age | Through study completion, an average of 6 months
  The age of a patient
Type of Cancer | Through study completion, an average of 6 months
  The type of cancer a patient has
Type of Treatment | Through study completion, an average of 6 months
  Type of cancer treatment a patient receives
Main Complaint | Through study completion, an average of 6 months
  Main complaint of ED visit
Physical parameters recorded during triage | Through study completion, an average of 6 months
  Physical parameters that are recorded during triage and are used in the prediction model
First Blood results | Through study completion, an average of 6 months
  The blood results that are recorded during triage and are used in the prediction model

CONTACTS AND LOCATIONS:
Overall Officials: Jason den Duijn, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No